CLINICAL TRIAL: NCT06228092
Title: A Blinded Randomized Study of Neostigmine/Glyco-pyrrolate 50 Mikrogram/kg or Sugammadex 2 mg/kg for Reversal of Neuromuscular Blockade in Elderly Patients (≥ 75 Years)
Brief Title: Neostigmine/Glyco-pyrrolate 50 Mikrogram/kg or Sugammadex 2 mg/kg for Reversal of Neuromuscular Blockade in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, MD, Ph.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-504230-21-00
Record Dates: First submitted 2023-11-03; First posted 2024-01-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Blockade, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Intervention Model Description: Randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neostigmine/glycopyrrolate group (Active Comparator): neostigmine/glycopyrrolate 50 mikrogr/kg
  Interventions: Drug: neostigmine/glycopyrrolate
- Sugammadex group (Active Comparator): Sugammadex 2 mg/kg
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: neostigmine/glycopyrrolate — Anesthesia personnel will administer the drug as a bolus over 5 seconds in an intravenous catheter upon conclusion of anaesthesia with a TOF within the range from TOF count of 2 to a TOF ratio < 0.60
  Other Names: Robinul-Neostigmin
  Arms: neostigmine/glycopyrrolate group
Drug: Sugammadex — Anesthesia personnel will administer the drug as a bolus over 5 seconds in an intravenous catheter upon conclusion of anaesthesia with a TOF within the range from TOF count of 2 to a TOF ratio < 0.60
  Other Names: Bridion
  Arms: Sugammadex group

SUMMARY:
The aim of this study is to determine the time to TOF ≥ 0.9 after either neostigmine/glycopyrrolate 50 mikrogr/kg or sugammadex 2 mg/kg in patients with age ≥ 75 years. The hypothesis of this study is that sugammadex 2 mg/kg provides a faster time to TOF ≥ 0.9 compared to neostigmine/glycopyrrolate 50 mikrogr/kg.

DETAILED DESCRIPTION:
Numbers of elderly patients requiring anesthesia and surgery are increasing, and as a group, elderly patients are at high risk of postoperative complications.

Although the use of neuromuscular blocking agents (NMBAs) to improve surgical condition are still debated, they are routinely administered in the clinical setting during anesthesia both to facilitate tracheal intubation and impair the surgical conditions. However, elderly patients administered NMBAs during anesthesia have an increased risk of postoperative residual neuromuscular block which is associated with more frequent episodes of hypoxemia, postoperative pulmonary complications, discomfort and longer hospital length of stay.

To prevent postoperative residual block it is strongly recommended to employ neuromuscular monitoring perioperatively, performed by train-of-four (TOF) stimulation, which enables the anesthetist to titrate the depth of block and to reverse the block if spontaneous recovery has not occurred upon conclusion of surgery.

It is possible to reverse rocuronium induced neuromuscular blockade with either neostigmine/glycopyrrolate (an acetylcholine esterase inhibitor) or sugammadex (a modified cyclodextrin). However, the optimal choice of reversal agent for rocuronium induced neuromuscular blockade in elderly patients is unknown. There is a need for studies investigating which reversal agent is optimal in elderly patients.

This randomized, parallel group trial will compare neostigmine/glycopyrrolate 50 mikrogr/kg or sugammadex 2 mg/kg for reversal of rocuronium induced blockade in elderly patients (≥ 75 years) undergoing robot surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 75 years old
2. Informed consent
3. Scheduled for robotic assisted laparoscopic surgery under general anesthesia with intubation and use of rocuronium during the entire operation
4. American Society of Anesthesiologists (ASA) physical status classification I to IV
5. Can read and understand Danish

Exclusion Criteria:

1. Known allergy to rocuronium, sugammadex or neostigmine/glycopyrrolate
2. Neuromuscular disease that may interfere with neuromuscular data
3. Severe renal impairment defined as eGFR < 30 ml/min
4. Indication for rapid sequence induction
5. Known intestinal or ureter obstruction
6. Known peritonitis

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Time to TOF > 0.9 | first TOF ratio ≥ 0.9 (time until complete recovery from effect of muscle relaxant) followed by a stable signal with a TOF ratio ≥ 0.9 for at least two minutes.
  time to TOF ≥ 0.9 after administration of either sugammadex or neostigmine/glycopyrrolate

SECONDARY OUTCOMES:
Residual muscular blockade | Assessed upon arrival at PACU, after 20 minutes at PACU and after 90 minutes at PACU
  Sign of residual muscular blockade defined as a composite (assessed upon arrival at PACU) of either:
  hand grip strength for 5 seconds; occurrence of double vision/blurred vision (yes/no); ability to track objects with eyes (follow finger of examiner) (yes/no); ability to sustain head lift for 5 seconds (yes/no); ability to protrude the tongue for 5 seconds (yes/no); tongue depressor test (prevent removal of a wooden tongue depressor from between the incisor teeth (yes/no); ability to open the eyes for 5 seconds (yes/no); ability to smile (yes/no); ability to speak (yes/no); occurrence of dysphagia/ swallowing impairment (ability to drink 20 ml of water) (yes/no); occurrence of upper airway obstruction; subjective symptoms of muscle weakness (whether the patient think a test was difficult to complete or uncomfortable to perform), recorded as normal (negative response) or impaired (positive response)

OTHER OUTCOMES:
Episodes of desaturation | During the period of the PACU stay
  Occurrence of episodes of desaturation defined as more than 3 minutes with spO2 < 88%.
New cardiac arrythmias | Within 180 minutes after administration of reversal agent
  Occurrence of new cardiac arrythmias (bradycardia or tachycardia defined as atrial fibrillation, atrial flutter, sinus tachycardia (>95 bpm), sinus bradycardia (<45 bpm))
Airway obstruction | During the period of the PACU stay
  Occurrence of upper airway obstruction
Reintubation | During the period of the PACU stay
  Occurrence of reintubation

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, MD, PhD, Study Chair — Rigshospitalet University of Copenhagen
Locations (3):
- Denmark (3):
  - Department of anaesthesia, Centre of Head and Orthopedics, Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Department of Pediatric and Obstetric Anaesthesia, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vested M, Wadland SS, Christensen MI, Creutzburg A, Madsen KPD, Tsuchiya EA, Madsen BG, Rovsing ML, Meyhoff CS, Lindelof K, Afshari A, Rasmussen LS. Neostigmine Versus Sugammadex for Reversal of Neuromuscular Blockade in Elderly Patients: A Blinded Randomised Study. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70160. doi: 10.1111/aas.70160. PMID 41307280

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT06228092/Prot_SAP_000.pdf